CLINICAL TRIAL: NCT05872880
Title: A Multicenter Prospective Real-world Study of TPExtreme Induced Chemotherapy Followed by Radical Surgery/Modified Radical Surgery and Radiotherapy in the Treatment of Locally Advanced Oral Squamous Cell Carcinoma.
Brief Title: TPExtreme Induced Chemotherapy Followed by Surgery and Radiotherapy in the Oral Carcinoma.
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Hunan Cancer Hospital (Other); The Second Hospital University of South China (Other)
Responsible Party: Sponsor
Other Study IDs: 202211261
Record Dates: First submitted 2023-02-08; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2022-11

CONDITIONS: Oral Squamous Cell Carcinoma; Locally Advanced Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TPExtreme induced chemotherapy was followed by modified radical surgery and radiotherapy: The effect was evaluated at three weeks after 2 cycles of TPExtreme(albumin-paclitaxel+cisplatin+cetuximab) induction chemotherapy according to the RECIST 1.1 guideline, lesion reduction by at least 50% can be included in our study. Patients choose modified radical surgery based on the tumor invasion scope after induction chemotherapy.
  In this group, the incisal margin was located 1~1.5cm outside the boundary of the residual tumor lesion after induced chemotherapy. At the same time, improved radical neck dissection was performed on both sides of the affected neck. Postoperative conventional radiotherapy(or chemoradiotherapy) was performed within 4 to 6 weeks after surgery.
  Interventions: Procedure: Modified radical surgery
- TPExtreme induced chemotherapy was followed by radical surgery and radiotherapy: The effect was evaluated at three weeks after 2 cycles of TPExtreme(albumin-paclitaxel+cisplatin+cetuximab) induction chemotherapy according to the RECIST 1.1 guideline, lesion reduction by at least 50% can be included in our study. Patients choose radical surgery based on the tumor invasion scope before induction chemotherapy.
  In this group, the incisal margin was located 1~1.5cm outside the boundary of the tumor lesion before induced chemotherapy. At the same time, radical neck dissection was performed on both sides of the affected neck. Postoperative conventional radiotherapy(or chemoradiotherapy) was performed within 4 to 6 weeks after surgery.
  Interventions: Procedure: Radical surgery

INTERVENTIONS:
Procedure: Modified radical surgery — The modified radical surgery was performed within 4 to 6 weeks after the end of the last chemotherapy, and local extended resection was performed according to the scope of the residual tumor lesions after induction therapy: the incisal margin was 1 to 1.5cm outside the boundary of the residual tumor lesions, and multi-point incisal rapid disease detection was performed intraoperatively to ensure negative incisal margin and complete resection of the residual tumor lesions. Under this premise, the surgical trauma should be minimized, and the organs and appearance of the patient should be preserved. For example, facial skin should not be penetrated, mandible should not be cut off, and tongue tissue should be preserved as much as possible. Direct suture or local tissue flap should be used to repair the defect during the operation. At the same time, improved radical neck dissection was performed on the affected side of the neck.
  Other Names: TPExtreme induced chemotherapy; radiotherapy
  Groups: TPExtreme induced chemotherapy was followed by modified radical surgery and radiotherapy
Procedure: Radical surgery — Radical surgery was performed within 4 to 6 weeks after the end of the last chemotherapy, and a wide range of radical surgical resection was performed according to the tumor scope before induction therapy: the incisal margin was 1 to 1.5cm outside the tumor boundary before induction, the lower lip and mandible could be incised if necessary, the facial skin could be excised, the mandibular bone segmentectomy was feasible, and pedicle or free skin (bone) flap was used to repair the defect. At the same time, improved radical neck dissection was performed on both sides of the affected neck.
  Other Names: TPExtreme induced chemotherapy; radiotherapy
  Groups: TPExtreme induced chemotherapy was followed by radical surgery and radiotherapy

SUMMARY:
Research shows that most oral cancer patients are already locally advanced when first diagnosed. Even after surgery and radiation, nearly half of patients develop recurrence or metastasis. Even in patients who survive, there is a serious decline in quality of life due to the after-effects of surgery and radiation. Many patients therefore refuse surgery and lose the treatment opportunity. Many studies at home and abroad have found that preoperative induction chemotherapy for locally advanced tumors can reduce tumor load, reduce tumor scope, eliminate distant micro metastases, reduce the risk of recurrence and metastasis, and improve organ preservation rate. It has been confirmed in many clinical studies and our clinical practice of oral cancer MDT(Multi-Disciplinary Treatment) that induction chemotherapy with TPExtreme protocol (cetuximab + albumin-paclitaxel + cisplatin) for patients with locally advanced oral cancer can significantly reduce the tumor with a good objective response, which can create good conditions for surgery. Therefore, for patients sensitive to induction chemotherapy, there are no authoritative guidelines and clinical studies to say what is the scope of surgery. One option is for the thoroughness of the tumor resection, which is still the same as the scope of the tumor before induction therapy, but the scope of the surgery is still large, and the damage to the patient's quality of life is also serious. The other option is to perform modified radical surgery according to the scope of residual tumor lesions after induction therapy, with less trauma and less damage to the quality of life. Postoperative radiotherapy (chemical) therapy is to reduce the risk of recurrence. Our preliminary clinical practice also shows that Patients sensitive to induction chemotherapy can obtain better survival rate and quality of life after comprehensive treatment including modified radical surgery. This treatment mode is feasible, but the overall efficacy evaluation needs further study. Therefore, in this real world prospective clinical study, patients with oral cancer sensitive to induction chemotherapy will be treated with modified radical surgery or traditional radical surgery in full compliance with the patient's wishes. Through clinical observation and follow-up statistics. To explore the effects of two treatment regimens on survival rate and quality of life in order to find the best treatment mode.

DETAILED DESCRIPTION:
Statistics showed that 65% of patients with oral cancer had been locally advanced when they were first diagnosed, and the tumor load was large. Even after radical surgical resection and radiotherapy, about 45% of patients with locally advanced oral cancer still have recurrence or metastasis, and the prognosis is poor. Even if the patients survive, due to the damage to tissues and organs caused by large-scale surgical excision, they often have a greater impact on the functions and appearance of the patients, such as chewing, swallowing, language, etc., the quality of life of the patients is generally poor and the medical costs are relatively high. Many studies at home and abroad have found that preoperative induction chemotherapy for advanced tumors can shrink tumor scope, eliminate distant micro metastases, reduce the risk of recurrence and metastasis, and improve organ preservation rate. It has been confirmed in many clinical practice that induction chemotherapy with TPExtreme protocol (cetuximab + albumin-paclitaxel + cisplatin) for patients with locally advanced oral cancer can significantly reduce the tumor volume with a good objective response rate (up to about 80%), which can create good conditions for surgery. The specific scheme was albumin paclitaxel 200mg/m2 D1; Cisplatin 75mg/m2, divided into 2-3 days; Cetuximab 400mg/m2 D1(250mg/m2 D8,D15), one cycle of treatment is 21 days, a total of 2 courses. However, for patients sensitive to induction chemotherapy, there has been no clear guideline on how to define the scope of surgical resection after tumor shrinkage or even disappearance, and there is also a lack of relevant clinical research to explore this. According to the RECIST 1.1 guideline for response evaluation criteria in solid tumors, equal or more than 50% reduction in lesion size can be included in this study. Patients fit the clinical trial criteria divide into two groups according to the patient's wishes. One group is radical surgery, patients receive surgery based on the tumor size before induction therapy, the other group is modified radical surgery who undergoes surgery based on the tumor size after induction therapy. Radical surgery is more extensive than modified radical surgery, and often requires mandibulectomy and internal fixation, as well as free flap transplantation to repair and reconstruct oral and maxillofacial defects, so it may need to use some special equipment. Such as titanium plate and titanium nail for internal fixation, microvascular anastomosis device, etc. However, modified radical surgery has a relatively small surgical range and is less likely to use the above devices. And during the operation, the incisal margin was 1~1.5cm outside the tumor boundary. If necessary, the lower lip and mandible could be incised, the facial skin could be excised, the mandibular bone could be segmental excision, and the defects could be repaired by pedicle or free skin (bone) flap. At the same time, improved radical neck dissection was performed on both sides of the affected neck. In operation, multiple incisal margin rapid disease examination was performed during the operation to ensure negative incisal margin and complete resection of the residual tumor lesion. Under this premise, minimize surgical trauma and preserve the patient's organs and appearance. Postoperative radiotherapy (or chemoradiotherapy) therapy to reduce the risk of recurrence. Postoperative radiotherapy was performed within 4-6 weeks after surgery. Linear accelerator/conformal intensity modulated radiotherapy was used for radiotherapy, and primary site radiotherapy was performed once a day, 5 times a week. The specific dose of radiotherapy is: PGTV(residue)：66-70Gy/30-33f(2-2.2Gy/f), PGTVtb(no residue):60-66Gy/30-33f(2-2.2Gy/f) , PGTVnd/ndtb：60-70Gy/30-33f(2-2.2Gy/f), high risk PTV：60Gy/30f(2Gy/f), low risk PTV：54Gy/30f(1.8Gy/f)。Our preliminary clinical practice showed that more and more patients with oral cancer tend to accept relatively less traumatic surgical programs, and patients sensitive to induction chemotherapy can obtain better survival rates and quality of life through modified radical surgery and postoperative adjuvant radiotherapy. This treatment mode is feasible, but the overall efficacy evaluation needs further study. Therefore, in this real world prospective clinical study, patients with oral squamous cell carcinoma sensitive to induction chemotherapy will be treated with modified radical surgery or traditional radical surgery in full compliance with the patient's wishes (without any biased intervention in the patient's clinical medical treatment). Through clinical observation and follow-up statistics. To explore the effects of two treatment regimens on survival rate and quality of life in order to find the best treatment mode.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG(Eastern Cooperative Oncology Group) score: 0~1.
2. New patients, confirmed by pathological biopsy for squamous cell carcinoma of the oral mucosa.
3. Tumor site: the tongue body, mouth floor, gums, buccal mucosa, after the hard palate, molar area.
4. TNM(Primary Tumor, Regional Node, Metastasis) staging (stage Ⅲ - Ⅳ B): T2-4bN0-3bM0.
5. After the assessment of tumor can be excised completely, or after the induction therapy may be removed completely.
6. can tolerate set by general treatment, no surgical contraindications, through the basin of chest CT + body Bone radionuclide scanning or PET-CT(Positron Emission Tomography / Computed Tomography) to rule out distant metastasis.
7. Pregnancy tests were performed in women of childbearing age (15-49 years old) within 7 days before treatment and the results were negative; Fertile male and female patients must consent to the use of effective contraceptive measures to ensure that during the trial and three months after withdrawal of pregnancy.
8. voluntarily signed informed consent and are willing and able to comply with the requirements of the study schedule follow-up, treatment, Laboratory testing and other research requirements.

Exclusion Criteria:

1. Have previously received relevant antitumor therapy, including chemotherapy, radiotherapy and immunotherapy.
2. Refused to sign the informed consent.
3. Patients who refuse to accept treatment options in clinical studies: patients who cannot get treatment to proceed smoothly; Patients unable to cooperate with regular follow-up due to psychological, social, family and geographical reasons.
4. Known to be allergic to the drugs that may be used to treat it.
5. For patients with poor general condition who cannot tolerate treatment. (Routine examination, such as three routine examinations, blood biochemical examination, electrocardiogram, chest radiograph, etc, to judge the general condition, when the results prompt HB(hemoglobin)<60g/L, WBC(white blood count)<3.0×10^9/L, PLT(platelet count)<80×10^9/L, Serum creatinine>133umol/L, it was considered that the general condition was poor and the treatment could not proceed smoothly, so conservative treatment was recommended)
6. Staging did not meet the inclusion criteria: patients with early clinical T1-2N0 oral cancer or patients with distant metastatic M1.
7. Assess patients who cannot be surgically resected, such as primary lesions or cervical metastases that invade vital structures such as the craniocerebral vital centers and carotid arteries.
8. Pregnant or lactating women (pregnancy tests should be considered for sexually active women of childbearing age).
9. Patients with past or current malignancies other than adequately treated non-melanoma skin cancer, cervical carcinoma in situ, and thyroid papillary carcinoma.
10. Participated in other clinical studies within the past 30 days.
11. Other conditions assessed by the researchers that could compromise patient safety or poor compliance, such as having a serious illness (including mental illness), severely abnormal test results, and other family or social high-risk risk factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1.From 18 to 65 years old; 2. The ECOG score is 0 to 1; 3. Newly diagnosed patients with locally advanced resectable/potentially resectable stage ⅲ-ⅳb oral mucosal squamous cell carcinoma (T1-2N1-3M0, T3-4bN0-3bM0).
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 60 months
  From the day of enrollment until treatment failure, death from any cause, or the last follow-up, the end point was the first occurrence.
Objective response rate | 60 months
  It refers to cases in which the tumor shrinks to complete and partial response after therapy.
Major partial response | 60 months
  The pathological reaction of the primary tumor after induction therapy was defined as the residual survival tumor ≤10%.

SECONDARY OUTCOMES:
Overall survival | 60 months
  From the day of enrollment until death from any cause or the last follow-up.
Locoregional failure-free survival | 60 months
  From the day of enrollment until local and/or regional recurrence or the last follow-up.
Distant failure-free survival | 60 months
  From the day of enrollment until distant metastasis or the last follow-up.

OTHER OUTCOMES:
Changes in patients' quality of life during treatment | 60 months
  Patients' quality of life was assessed using the head and neck specific module First Edition (H&N35) of the Quality of Life Questionnaire - Core 30 Modules third Edition (QLQ-C30) developed by the European Organization for Research and Treatment of Cancer (EORTC). The questionnaire was scored on a scale of 0 to 100, with higher scores indicating better functioning or quality of life, or heavier symptom load.
Assessment of toxicity and general conditions during and after treatment | 60 months
  Acute subjective toxic reactions to chemoradiotherapy: According to NCI-CTC 5.0 criteria, subjective toxic reactions were evaluated once per cycle during chemotherapy and once per week during radiotherapy. Objective acute toxic reactions of chemoraochemotherapy: According to the NCI-CTC 5.0 standard, blood routine and biochemical examination were performed before each course of chemotherapy, and once on the 3rd and 7th day after each course of chemotherapy and 1 day before the next course of chemotherapy. Objective toxic reactions were assessed by weekly blood draws during radiotherapy. The results with higher grades are taken as the comprehensive results. When the grade of adverse event is greater than or equal to grade 3, the patient is considered unable to continue treatment successfully.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No